CLINICAL TRIAL: NCT02739425
Title: SMART Study: Sentimag Along With Routine Technique in Detection of Sentinel Node Biopsy
Brief Title: The Efficacy of Sentimag in Detection of Sentinel Node Biopsy
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Collaborators: Sysmex Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015SUR79
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; Sentinel Node
Keywords: Sentinel lymph node biopsy (SLNB); Superparamagnetic iron oxide (SPIO) tracer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Standard Procedure plus use of sentimag (Other): Detection of the nodes carried out using the gamma probe and also the sentimag - all patients receive both diagnostic interventions
  Interventions: Device: Sentimag Device

INTERVENTIONS:
Device: Sentimag Device — The programme will compare the Sentimag with the conventional sentinel lymph node detection with radioactive tracer combined with blue dye (in centres using the combined technique) and thereby determine whether the new technique is equivalent to the standard technique for SLNB

SUMMARY:
The aim of this study is to evaluate the Sentimag/Sienna+ System (Sentimag®) in clinical routine practice. On the one hand this allows evaluation of the equivalence of the two techniques. On the other hand this ensures that patients do not experience any possible disadvantages by participating. The hypothesis behind this evaluation is that Sentimag is as efficient as conventional sentinel node mapping.

The programme will compare the Sentimag® with the conventional sentinel lymph node detection with radioactive tracer combined with blue dye (in centres using the combined technique) and thereby determine whether the new technique is equivalent to the standard technique for SLNB.

DETAILED DESCRIPTION:
Sentinel lymph node biopsy (SLNB) is now the standard technique used in breast cancer patients with a clinically and radiologically negative axilla. SLNB for breast cancer was introduced in the 1990s3 and it significantly reduces the morbidity associated with axillary node dissection (ALND) including lymphedema, seroma, numbness, wound infection, reduced shoulder motility, and chronic pain.2 The gold standard for sentinel node detection is the 'combined technique'; using both blue dye and radioisotope injection. After allowing both radioisotope and blue dye to localize in the lymphatic system, the clinician uses a 'gamma probe' (a handheld scintillation counter) to locate the SLNs. The blue dye assists in localisation post-incision, with lymph nodes that are blue and/or radioactive are judged as 'SLNs' and excised. Some centres use either radioisotope or blue dye alone. Although detection rates are lower, they can still reach satisfying values in experienced centres.

The use of radioisotope exposes patients and healthcare workers to radiation, is heavily controlled by legislation (both on the specific training for operators and subsequent disposal of surgical waste), and provides poor pre-operative imaging. As a result, many centres have stopped undertaking routine pre-operative lymphoscintigraphy. There is thus a clinical need to develop new techniques for detecting sentinel nodes without these drawbacks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary breast cancer scheduled for Sentinel node biopsy;
* Patients who are clinically and radiologically node negative;.
* Patients aged ≥18 years at time of consent
* Patients are able and willing to give informed consent
* Ability and willingness to undertake all scheduled visits and assessments

Exclusion Criteria:

* Patients who are currently Pregnantcy or lactatingon;
* Patients with metastatic cancer;
* Subject has a known hypersensitivity to blue dye;
* Patients with intolerance or hypersensitivity to iron oxide or dextran compounds;, or to Sienna+
* Patients who have iron overload disease;
* Patients who has a pacemaker or other implantable device in the chest wall or shoulder;
* Previous axilla surgery, or impaired lymphatic function
* Subject is deprived of liberty or under guardianship
* Subject is indicated or scheduled for post-operative MRI investigation of the breast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Proportion of successful sentinel node biopsies (SLNB, detection rate per patient) with either the magnetic or the standard technique | 6 Months

SECONDARY OUTCOMES:
Detection rate per node | 6 Months
Malignancy rate: proportion of nodes and patients with a malignant result in the definite pathological analysis. | 6 Months
Concordance rate: proportion of successful labelling with the standard and new technique per patient and per node | 6 Months
Malignancy concordance: proportion of successful labelling with the standard and new technique per malignancy positive patients and nodes | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Raghavan Vidya, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided